CLINICAL TRIAL: NCT03935620
Title: Delivering Early Intervention to Children With Down Syndrome Through Telemedicine
Brief Title: Delivering Early Intervention to Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Emily Quinn, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018508
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A single case multiple-baseline across behaviors (i.e., EMT strategies) design-replicated across ten caregiver-child dyads will be used to evaluate the effect of implementing EMT via telepractice on parent's EMT strategy usage and concomitant increases in child communication. Within each design there will be three potential demonstrations of effect and three potential replications across participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMT (Experimental): After a period of stable baseline performance (3 to 5 sessions) for parents and children the interventionists will apply the EMT Language Intervention.
  Interventions: Behavioral: Enhanced Milieu teaching

INTERVENTIONS:
Behavioral: Enhanced Milieu teaching — Enhanced Milieu Teaching (EMT) an evidence-based, naturalistic language intervention that has been optimized to address the specific language and communication deficits associated with DS. EMT is a parent-implemented intervention that involves home-visits during which clinicians teach parents to support their child learning language during typical parent-child interactions at home (play with toys, music, book reading, and snack time). Clinicians follow an evidence-based instructional framework called "Teach-Model-Coach-Review" to teach parents language support strategies.

SUMMARY:
Children with Down syndrome (DS) are at risk for significant language and communication impairments. Enhancing the service delivery of early intervention for children with DS is a key research and policy issue given the prevalence and detrimental effects of persistent language impairments. Using a telemedicine approach allows clinicians to provide evidence-based treatment to families from a wide geographic area in Oregon who may not otherwise have access to a language intervention specialized for children with DS. Our innovative project involves the creation of a new treatment optimized for children with DS, as it will be the first study that translates an existing evidence-based language intervention-Enhanced Milieu Teaching (EMT) into a telemedicine model. The goal of this study is to examine whether a telemedicine approach is effective for training parents to implement EMT language support strategies and whether changes in parent behavior are associated with child communication and language growth. The investigators will pilot the telemedicine initiative to provide early intervention services to ten children with DS (aged 18- 48 months) and their families who live in rural and /or under-served areas of Oregon. The investigators will use single-case research design methodology to pilot this intervention research. The investigators will use secure video-teleconferencing technology to provide EMT. Clinicians will provide EMT to parents through interactive coaching, teaching them how to foster their children's social communication and language skills. Outcomes will focus on parents' use of language support strategies and children's social communication and language skills. Delivering early intervention to children with DS and providing parent-training at a distance using a telemedicine approach has the potential to transform the delivery of early language interventions for children with DS. Results of this study will directly inform the development and refinement of language interventions for young children with DS.

DETAILED DESCRIPTION:
1. Aim 1: To examine the effect of using a telemedicine service delivery model to teach parents of children with DS to use EMT language support strategies. The investigators hypothesize that parents will learn to use EMT language support strategies from the personalized instruction provided during 36 intervention sessions.
2. Aim 2: To examine the effect of delivering EMT using a telemedicine service delivery model to improve the spoken language and social communication skills of children with DS. The investigators hypothesize that improvements in child communication and language skills will result from increasing parents' use of EMT language support strategies during everyday parent-child interactions such as play with toys, singing songs, book reading, and mealtimes.

ELIGIBILITY:
Inclusion Criteria:

* child age between 18 and 36 months
* developmental age of 9 months as measured on the Visual Reception Scale of the Mullen Scales of Early Learning (MSEL; Mullen, 1995)
* primary diagnosis of Down syndrome as indicated in medical history,
* secondary diagnosis of language delay as measured by a score of at least 1.33 SD below the mean on the Preschool Language Scales -5th Edition (PLS-5; Zimmerman, Steiner, & Evatt-Pond, 2011),
* hearing (with or without amplification) reported at 25dB HL or better confirmed by audiological testing, or medical record.

Exclusion Criteria:

* concomitant sensory impairments (e.g., hearing impairment, blindness), and
* symptoms of autism spectrum disorder as measured by a result indicating "high risk" for autism (e.g., scores of 8 or higher) on the Modified Checklist for Autism In Toddlers-Revised with Follow-up (MCHAT-R/F Robins, Fein & Barton, 2009).

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Between Session Change:Number of EMT Strategies Used by Parents During Parent-Child Interaction | Assessed 1-2 times per week for 3- 4 months.
  Observational measure coded from video-recordings of a 15 minute caregiver-child interaction. 10 minutes of play and toys and 5 minutes of a home routine. Changes in the number of different EMT strategies used by parents will be quantified.

SECONDARY OUTCOMES:
Between Session Change: Rate of Symbolic Communication During Parent-Child Interaction | Assessed 1-2 times per week for 3-4 months.
  Observational measure coded from video-recordings of a 15 minute caregiver-child interaction. 10 minutes of play and toys and 5 minutes of a home routine.
Communication Matrix Scores | Assessed at T00 (Study Entry) and T01 (3- 4 months post intervention).
  Total score on an assessment of early expressive communication skills.
Between Session Change: Number of Different Words Expressed During Parent-Child Interaction | Assessed 1-2 times per week for 3-4 months.
  Observational measure coded from video-recordings of a 15 minute caregiver-child interaction. 10 minutes of play and toys and 5 minutes of a home routine.

CONTACTS AND LOCATIONS:
Overall Officials: Emily D Quinn, Ph.D, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States